CLINICAL TRIAL: NCT01536184
Title: Evaluating the Effectiveness of an Attachment-Focused Intervention in Preschool Children With Fetal Alcohol Spectrum Disorder (FASD) or At-risk for FASD: A Randomized Controlled Field Trial
Brief Title: Evaluating the Effectiveness of an Attachment-Focused Intervention in Preschool Children With FASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Ana Hanlon-Dearman, Developmental Pediatrician, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2012:015
Record Dates: First submitted 2012-02-09; First posted 2012-02-20 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Fetal Alcohol Spectrum Disorder; Attachment Disorders
Keywords: Fetal Alcohol Spectrum Disorder; FASD
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receives COS Intervention (Experimental): Circle of Security (COS) Family Intervention (B. Marvin model) is a community based, visually supported, individualized attachment protocol appropriate for use with preschoolers and children and their parents/caregivers. The goals of the intervention include increasing caregiver sensitivity and appropriate responsiveness to their child through increasing their capacity to recognize and understand their child's cues, and increasing caregiver self-reflection on their own caregiving behaviour. The protocol itself involves a series of activities and repeated videotaped interactions between the child and their caregiver which are reviewed by the therapist who has established themselves with the caregiver as a secure base from which the attachment relationship may be explored.
  Interventions: Behavioral: Circle of Security (COS)
- Control Group-Regular FASD Services (No Intervention): Regular FASD Services include general information on Fetal Alcohol Spectrum Disorder (FASD) with general behavioural management strategies and parental supports.

INTERVENTIONS:
Behavioral: Circle of Security (COS) — COS is a community based, visually supported, individualized attachment protocol appropriate for use with preschoolers and children and their parents/caregivers. It is based on attachment theory of John Bowlby and Mary Ainsworth and integrates neuroscientific principles of emotional regulation and attachment. The protocol contains both educational and therapeutic components. The goals of the intervention include increasing caregiver sensitivity and appropriate responsiveness to their child through increasing their capacity to recognize and understand their child's cues, and increasing caregiver self-reflection on their own caregiving behaviour.
  Other Names: Attachment Intervention
  Arms: Receives COS Intervention

SUMMARY:
Study Summary: This study is being conducted in order to rigorously evaluate the real-world effectiveness of a publicly-funded, home-based, attachment-focused intervention Circle of Security (COS) Family Intervention Model (Marvin) in improving caregiving and child outcomes in families who have children with Fetal Alcohol Spectrum Disorder (FASD) or who are at-risk for FASD, as delivered under routine practice conditions.

Hypothesis: At post-test (after 36 sessions and 3-month follow-up), compared to a wait-list control group receiving standard services, the treatment group receiving COS will show greater improvement in caregiver behaviour, as well as child emotional and behavioural outcomes.

DETAILED DESCRIPTION:
See Arms and Intervention

ELIGIBILITY:
Inclusion Criteria:

* Two criteria must be present for a family (caregiver-child dyad) to be included in the COS component of the FASD Outreach Program and its evaluation:

  * the child was exposed to alcohol prenatally and has been clinically evaluated using the Canadian FASD diagnostic guidelines as having Fetal Alcohol Syndrome (FAS), Partial Fetal Alcohol Syndrome (PFAS), Alcohol Related Neurodevelopmental Disorder (ARND), or is considered "at risk" for FASD based on their confirmed history of prenatal alcohol exposure and clinical multidisciplinary assessment; and
  * evidence of disrupted caregiver behaviours or problems in the caregiver-child interaction as identified through a screening process consisting of clinical judgment and the SBSH procedure.

Exclusion Criteria:

* children from foster families who have experienced more than 2 placements in the last six months,
* children who have an Autism diagnosis,
* children with a developmental quotient less than 50,
* children with sensory impairments (hearing or sight impaired), and
* children who are already involved in New Directions' 'Self Regulation Therapy Project'.

Children who have parents who are clinically depressed, whose parents have substance abuse or domestic violence issues, or whose parents display a narcissistic devaluation personality trait based on initial clinical evaluation, will also be excluded from study eligibility.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Hanlon-Dearman, M.D., Principal Investigator — University of Manitoba; FASD Outreach, Study Chair — Family Services and Housing, Province of Manitoba; Healthy Child Manitoba Office, Study Chair — Government of Manitoba
Locations (1):
- FASD Outreach Program, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The population studied were families with preschool children with FASD or PAE who were referred to the provincial FASD Outreach program or the FASD Family Support, Education and Counselling Program, a program of New Directions,between January 2011 - December 2013. The age range of children in the FASD Outreach Program is between 2 to 5 years old.
Groups:
- Receives COS Intervention: Circle of Security (COS) Family Intervention (B. Marvin model) is a community based, visually supported, individualized attachment protocol appropriate for use with preschoolers and children and their parents/caregivers. The goals of the intervention include increasing caregiver sensitivity and appropriate responsiveness to their child through increasing their capacity to recognize and understand their child's cues, and increasing caregiver self-reflection on their own caregiving behaviour. The protocol itself involves a series of activities and repeated videotaped interactions between the child and their caregiver which are reviewed by the therapist who has established themselves with the caregiver as a secure base from which the attachment relationship may be explored.
  Circle of Security (COS): COS is a community based, visually supported, individualized attachment protocol appropriate for use with preschoolers and children and their parents/caregivers. It is based on attachment
Period: Overall Study
Arm/Group | Receives COS Intervention | Control Group-Regular FASD Services
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Receives COS Intervention | Control Group-Regular FASD Services | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Full Range); unit: years] | 4.1 [2 to 5] | NA [NA to NA] — Specific age data not collected by the community therapists. | 4.1 [2 to 5]
Age, Customized [Number; unit: Participants]
  Less than or equal to 5 years old | 8 | 4 | 12
  Greater than 5 years old | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Attachment Classification
Description: Attachment classified using Ainsworth's Strange Situation protocol: Secure, Anxious-Insecure, Anxious-Avoidant, Avoidant, Disorganized.
Time Frame: Administered 3 times: at baseline (pretest), 9 months (postest), 12 months (followup)
Population: Number of participants analyzed Receives COS Intervention Pretest= 8; Post-test=3; Follow-up=4 Control Group Pretest=4; Post-test=1; Follow-up=1
Measure: Number; unit: participants
Arm/Group | Receives COS Intervention | Control Group-Regular FASD Services
Number analyzed (Participants) | 8 | 4
participants
  Secure (pretest) | 0 | 0
  Anxious-Insecure (pretest) | 0 | 0
  Anxious-Avoidant (pretest) | 0 | 0
  Avoidant (pretest) | 3 | 0
  Disordered (pretest) | 5 | 4
  Secure (post test) | 1 | 0
  Anxious-Insecure (post test) | 0 | 0
  Anxious-Avoidant (post test) | 0 | 0
  Avoidant (post test) | 0 | 0
  Disordered (post test) | 2 | 1
  Secure (followup) | 1 | 0
  Anxioius-Insecure (followup) | 0 | 0
  Anxious-Avoidant (followup) | 0 | 0
  Avoidant (followup) | 0 | 0
  Disordered (followup) | 3 | 1

2. Secondary Outcome: The Parenting Scale (TPS)
Description: A self-report measure of dysfunctional parenting practices including laxness, over-reactivity, and verbosity. The scale has good internal consistency and test-restest reliability and scores are consistent with other measures of dysfunctional discipline and child misbehaviour.
  Each subscale score, ranges from 1 to 7; for each subscale (Laxness, Overreactivity, Verbosity) lower values indicate a lower degree of self-perceived ineffective parenting behaviors and higher values indicate a greater degree of self perceived ineffective parenting behaviours. The total score is calculated from a combination of each subscale and also ranges from 1 to 7, reflecting the degree of ineffective parenting behaviours across all categories with lower values indicate a lower degree of self-perceived ineffective parenting behaviors and higher values indicate a greater degree of self perceived ineffective parenting behaviours.
Time Frame: Administered 3 times: at baseline (pretest), 9 months (postest), 12 months (followup)
Population: Number of Participants Analyzed Receives COS Intervention Pretest= 8; Post-test=6; Follow-up=5 Control Group Pretest=4; Post-test=2; Follow-up=2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receives COS Intervention | Control Group-Regular FASD Services
Number analyzed (Participants) | 8 | 4
units on a scale
  TPS Total (pretest) | 4.08 [2.57 to 4.43] | 2.3 [1.71 to 3.13]
  TPS Total (post test) | 2.97 [2.4 to 4.07] | 3.27 [3.17 to 3.37]
  TPS Total (followup) | 2.67 [1.87 to 3.33] | 2.6 [2.03 to 3.17]
  TPS Laxness (pretest) | 3.22 [1.82 to 5.55] | 2.22 [1.56 to 4.55]
  TPS Laxness (post test) | 2.97 [1.81 to 5.0] | 3.14 [3.11 to 3.18]
  TPS Laxness (followup) | 2.47 [2.0 to 3.36] | 2.46 [1.91 to 3.0]
  TPS Overreactivity (pretest) | 2.39 [1.9 to 3.2] | 1.65 [1.2 to 2.2]
  TPS Overreactivity (post test) | 2.18 [1.8 to 2.6] | 2.53 [2.25 to 2.8]
  TPS Overreactivity (follow up) | 2.46 [1.5 to 3.5] | 1.85 [1.7 to 2.0]
  TPS Verbosity (pretest) | 3.54 [1.86 to 4.43] | 2.80 [2.0 to 4.0]
  TPS Verbosity (post test) | 3.56 [3.0 to 4.86] | 3.52 [3.17 to 3.86]
  TPS Verbosity (follow up) | 3.11 [2.14 to 4.29] | 3.36 [2.71 to 4.0]

3. Secondary Outcome: The Parenting Stress Index (PSI)
Description: A parent-report questionnaire of parental stress reflecting parent-child interaction style and difficult child behaviour. There are two main domain scores, a Child Domain Score and Parent Domain Score from which a Total Stress Score is calculated.
  Child and Parent Domain raw scores combine to form a Total Stress raw score. Higher scores for each item indicate a higher degree of negative attributes in the given scale while lower scores indicate lower relationship stress and a greater sense of enjoyment in the relationship.
  Items include:
  Defensive Responding (DR) Score range 7-35 Parental Distress (PD) Score range 12-60 Parent-Child Dysfunctional Interaction (PCDI) Score range 12-60 Difficult Child (DC) Score range 12-60 PSI Total Stress Score range 36-180
Time Frame: Administered 3 times: at baseline (pretest), 9 months (postest), 12 months (followup)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receives COS Intervention | Control Group-Regular FASD Services
Number analyzed (Participants) | 8 | 4
units on a scale
  DR (pretest) n=8, n=4 | 25.13 [11 to 34] | 14.25 [10 to 19]
  DR (post test) n=6, 1 | 15.66 [12 to 22] | 16 [16 to 16]
  DR (followup) n=5, n=2 | 19 [9 to 30] | 18 [17 to 19]
  PD (pretest) n=8, n=4 | 42.75 [17 to 57] | 24 [17 to 31]
  PD (post test) n=6, n=1 | 27 [20 to 38] | 29 [29 to 29]
  PD (followup) n=5, n=2 | 33.4 [14 to 52] | 30.5 [30 to 31]
  PCDI (pretest) n=8, n=4 | 37.5 [22 to 50] | 24.5 [16 to 33]
  PCDI (post test) n=6, n=1 | 25.66 [21 to 31] | 31 [31 to 31]
  PCDI (followup) n=5, n=2 | 27.8 [14 to 43] | 24 [19 to 29]
  DC (pretest) n=8, n=4 | 35.75 [28 to 46] | 40.75 [28 to 53]
  DC (post test) n=6, n=1 | 33.66 [20 to 44] | 56 [56 to 56]
  DC (followup) n=5, n=2 | 35.4 [25 to 42] | 42 [34 to 50]
  PSI total Stress (pretest) n=8, n=4 | 116 [89 to 144] | 89.25 [74 to 111]
  PSI total Stress (post test) n=6, n=1 | 86.33 [74 to 103] | 116 [116 to 116]
  PSI total Stress (followup) n=5, n=2 | 96.6 [53 to 128] | 96.5 [83 to 110]

4. Secondary Outcome: The Depression Anxiety Stress Scale (DASS)
Description: A self-report measure of depression, anxiety, and stress. The scales of the DASS show high internal consistency and produce meaningful discriminations in different settings, and are appropriate for measuring the emotional states of caregivers over time.
  The score for each item ranges from 0 to 3, where 0 indicates "did not apply to me at all" and 3 indicates "applied to me very much, or most of the time". The individual items are combined using a scoring template into measures of Depression (D), Anxiety (A), and Stress (S). Depression is scored out of 28 where 0-9 is normal and 10-28 reflect mild, moderate, and severe degrees of depression. Anxiety is scored out of 20 where 0-7 is normal and 8-20 reflect mild, moderate, and severe degrees of anxiety. Stress is scored out of 34 where 0-14 is normal and 15-34 reflect mild, moderate, and severe degrees of stress.
Time Frame: Administered 3 times: at baseline (pretest), 9 months (postest), 12 months (followup)
Population: Receives COS Intervention Pretest= 8; Post-test=6; Follow-up=5 Control Group Pretest=4; Post-test=2; Follow-up=2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receives COS Intervention | Control Group-Regular FASD Services
Number analyzed (Participants) | 8 | 4
units on a scale
  DASS-D (pretest) | 2.63 [0 to 13] | 1 [0 to 2]
  DASS-D (post test) | 3.33 [1 to 7] | 0 [0 to 0]
  DASS-D (followup) | 5.2 [0 to 17] | 0 [0 to 0]
  DASS-A (pretest) | 4.13 [0 to 11] | 0.5 [0 to 2]
  DASS-A (post test) | 4.5 [0 to 9] | 0 [0 to 0]
  DASS-A (followup) | 4 [0 to 16] | 0 [0 to 0]
  DASS-S (pretest) | 7.63 [2 to 19] | 3 [0 to 5]
  DASS-S (post test) | 6.17 [1 to 11] | 4.5 [0 to 9]
  DASS-S (followup) | 9 [2 to 18] | 2 [0 to 4]

5. Secondary Outcome: The Strengths and Difficulties Questionnaire SDQ
Description: The Emotional Symptoms (SDQ-ES), Conduct Problems (SDQ-CP), Hyperactivity (SDQ-HA), Peer Problems (SDQ-PP), and Prosocial (SDQ-PS) Scales each range from 0-10 Higher values in (ES, CP, HA, and PP) indicate a greater degree of abnormal behavior; low values indicate more normative behavior. For the PS scale, higher values indicate greater strengths in prosocial behaviour and lower values indicate more difficulties with prosocial behavior. A Total Difficulties Score ranges from 0 to 40 with higher scores reflecting higher levels of behavioral difficulty. The Total Impact Supplement Score (Total IS) ranges from 0 to 10 with higher values indicating greater behavioral difficulty and social impairment.
Time Frame: Administered 3 times: at baseline (pretest), 9 months (postest), 12 months (followup)
Population: Please see category specific n values below.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receives COS Intervention | Control Group-Regular FASD Services
Number analyzed (Participants) | 8 | 4
units on a scale
  SDQ-ES (pretest) n=7, n=4 | 2.86 [2 to 4] | 4.5 [2 to 7]
  SDQ-ES (post test) n=6, n=1 | 4.33 [2 to 8] | 3 [3 to 3]
  SDQ-ES (followup) n=5, n=2 | 3.8 [1 to 4] | 3 [1 to 3]
  SDQ-CP (pretest) n=5, n=4 | 5 [1 to 6] | 4.5 [1 to 8]
  SDQ-CP (post test) n=6, n=1 | 3.66 [0 to 7] | 7 [7 to 7]
  SDQ-CP (followup) n=5, n=2 | 4.8 [3 to 7] | 4 [1 to 7]
  SDQ-HA (pretest)n=6, n=4 | 8.17 [5 to 10] | 8 [6 to 10]
  SDQ-HA (post test) n=6, n=1 | 6.66 [4 to 10] | 9 [9 to 9]
  SDQ-HA (followup) n=5, n=2 | 7.8 [5 to 10] | 6.5 [5 to 8]
  SDQ- PP (pretest) n=7, n=4 | 3 [0 to 7] | 4 [3 to 5]
  SDQ- PP (post test)n=6, n=1 | 3.33 [1 to 5] | 6 [6 to 6]
  SDQ- PP (followup)n= 5, n=2 | 2.8 [1 to 4] | 3 [2 to 4]
  SDQ-PS (pretest) n=7, n=4 | 5.86 [4 to 7] | 6 [4 to 8]
  SDQ-PS (post test) n=6, n=1 | 6.66 [4 to 9] | 5 [5 to 5]
  SDQ-PS (followup) n=5, n=2 | 6.2 [6 to 8] | 7 [5 to 9]
  Total SDQ (pretest)n=7, n=4 | 18.71 [14 to 27] | 21 [15 to 25]
  Total SDQ (post test)n=6, n=1 | 18 [14 to 28] | 25 [25 to 25]
  Total SDQ (followup) n=5, n=2 | 19.2 [9 to 22] | 16 [10 to 22]
  Total IS (pretest) n=7, n=4 | 4.43 [1 to 8] | 5.5 [2 to 10]
  Total IS (post test) n=6, n=1 | 2.12 [0 to 5] | 10 [10 to 10]
  Total IS (followup)n=5, n=0 | 3.4 [2 to 7] | NA [NA to NA] — No data could be collected for this test as participant did not attend assessment

ADVERSE EVENTS:
Description: Adverse events were not assessed.
Arm/Group | Receives COS Intervention | Control Group-Regular FASD Services
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
While we set out to conduct an RCT to evaluate the effectiveness of COS delivered in a home-visiting model vs. a behavioral TAU intervention, the limitations we faced did not allow for this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No